CLINICAL TRIAL: NCT06579898
Title: The Effect of Progressive Resistance Exercise Training (PRET) on Cardiovascular Risk Factors in Adults With ID.
Brief Title: The Effect of Progressive Resistance Exercise Training (PRET) on CVRF in Adults With ID.
Acronym: PRET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Kirsten de Oude MSc, Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTR NL8382
Record Dates: First submitted 2024-03-07; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Hypercholesterolemia; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Hypercholesterolemia; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRET (Experimental): All participants participate in a progressive resistance exercise training programme for 24 weeks.
  Interventions: Other: Progressive resistance exercise training

INTERVENTIONS:
Other: Progressive resistance exercise training — A 24-week progressive strength training programme (PRET). Divided into 4 mesocycles in which the intensity of training is built up from 60% 1RM- 80% 1RM. Training is carried out twice a week under the guidance of a physiotherapist or exercise instructor.

SUMMARY:
Thanks to improved healthcare, the life expectancy of people with ID is increasing and is approaching that of the general population. Several studies have shown that most cardiovascular disease (CVRF) risk factors are as common or even more common in people with ID than in the general population. The guidelines of the American College of Sport Medicine (ACSM) state that a resistance training (RT) programme can can effectively reduce CVRF if performed at a high intensity. A secondary benefit of RT is the increase in muscle strength and muscle mass that can reduce and can improve the ability to perform activities of daily living (ADL), also two common problems in people with ID.

DETAILED DESCRIPTION:
This study has a repeated time series design with one study group. The study period will last one year and is divided into a 12-week baseline period, a 24-week intervention period (PRET programme), and a 12-week follow-up period. The PRET programme will take 24 weeks and consists of two sessions per week, with at least 48 hours between the sessions. The intervention will be led by experienced physiotherapists and physical activity instructors employed by the care providers. All instructors take part in a training prior to the study. In this training, the intervention protocol and exercises will be discussed and practiced ensuring that the intervention is delivered according to the protocol. Every session consists of seven exercises (RESID) to train all large muscle groups. The programme is in accordance with the ACSM guidelines and characterised by four mesocycles. Each mesocycle consists of six weeks of training. After each mesocycle the training intensity will increase gradually, and within each mesocycle the weights will be adjusted in a way that the intensity remains equal. Training intensity will be measured by the percentage of the heaviest load one can lift for one repetition (% of 1RM). In the first mesocycle, participants are introduced to the resistance exercises and familiarised to the training protocol. They will learn to perform the exercises safely and with good posture. During mesocycles 2, 3, and 4, the number of repetitions will be gradually decreased while the training intensity will be gradually increased until vigorous intensity is reached in the fourth mesocycle (80% of 1RM). The resting time between sets will depend on the training intensity and varies between 30 seconds and 2 minutes. The instructors will register attendance, training intensity, performed number of sets and repetitions, and the weights used for each exercise in a log.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older;
* living in a residential facility or receiving care from one of the participating care providers;
* diagnosed with mild (IQ = 50-69) or moderate (IQ = 35-49) ID;
* diagnosed with metabolic syndrome, or at least two of the following CVRF: hypertension, hypercholesterolemia, diabetes mellitus type 2, or obesity.
* participants must be able to walk independently and able to follow instructions on posture and performance for good execution of the exercises

Exclusion criteria:

not able to follow instructions or physical limitations interfering with participation in training programme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Glycated Haemoglobin | through study completion, an average of 1 year
  mmol/mol, Outcome is measured with blood samples and analysed in a laboratory of ErasmusMC
Systolic blood pressure | through study completion, an average of 1 year
  mm/Hg, Blood pressure is measured with a digital blood pressure device
LDL cholesterol | through study completion, an average of 1 year
  mmol/L, Outcome is measured with blood samples and analysed in a laboratory of ErasmusMC
Waist-hip ratio | through study completion, an average of 1 year
  cm, Waist-hip ratio is calculated after measuring waist circumference and hip circumference with a flexible tape measure.

SECONDARY OUTCOMES:
Triglycerides | through study completion, an average of 1 year
  mmol/L, Outcome is measured with blood samples and analysed in a laboratory of ErasmusMC
HDL cholesterol | through study completion, an average of 1 year
  mmol/L, Outcome is measured with blood samples and analysed in a laboratory of ErasmusMC
Total cholesterol | through study completion, an average of 1 year
  mmol/L, Outcome is measured with blood samples and analysed in a laboratory of ErasmusMC
Glucose | through study completion, an average of 1 year
  mmol/L, Outcome is measured with blood samples and analysed in a laboratory of ErasmusMC
Muscle strength | through study completion, an average of 1 year
  kg, Muscle strength is measured with handgrip strength, 30 second chair stand and 5 times chair stand
Muscle mass | through study completion, an average of 1 year
  kg, Muscle mass is measured with a bio electrical impedance device
(I)ADL questionnaire | through study completion, an average of 1 year
  (I)ADL is measured with a questionnaire, which is filled in by proxy
Fall incidents | through study completion, an average of 1 year
  Falls are reported during baseline and follow up with a calandar filled in by proxy
ABC questionnaire | through study completion, an average of 1 year
  Behavioural issues is measured with the ABC questionnaire, which is filled in by proxy

CONTACTS AND LOCATIONS:
Overall Officials: Alyt Oppewal, Dr, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - Amarant, Tilburg, North Brabant
  - Abrona, Huis Ter Heide, South Holland
  - Ipse de Bruggen, Zoetermeer, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Study protocol has been published. Further information can be requested.
Supporting Information: Study Protocol
Time Frame: Study Protocol is available Elbers RG, de Oude KI, Kastanidis T, Maes-Festen DAM, Oppewal A. The Effect of Progressive Resistance Exercise Training on Cardiovascular Risk Factors in People with Intellectual Disabilities: A Study Protocol. Int J Environ Res Public Health. 2022 Dec 8;19(24):16438. doi: 10.3390/ijerph192416438. PMID: 36554319; PMCID: PMC9778210.
Access Criteria: Open access